CLINICAL TRIAL: NCT04095546
Title: Epigenetic Changes in Psychotherapy of Adolescents With Borderline Personality Pathology
Status: Withdrawn | Type: Observational
Why Stopped: personal changes in study team
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Leading House for the Latin American Region (Seed Money Grant SMG 1730) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-00658; pk19Zimmermann
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Borderline Personality Disorder (BPD)
Keywords: epigenetic changes; Psychotherapy; epigenetic regulation; methylation patterns; change in methylation of genes; FKBP5 gene
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: routine psychotherapy for Borderline Personality Disorder (BPD) — Routine psychotherapy as treatment for patients with Borderline Personality Disorder

SUMMARY:
The link between epigenetic changes as an effect of psychotherapy has been investigated recently. Genes investigated in these studies were brain-derived neurotrophic factor (BDNF), NR3C1, FKBP51, MAOA and GLUT1. Change in methylation of these genes could be a biomolecular mechanism of psychotherapy induced changes. This study project aims at providing evidence for a biological mechanism of personality disorder interventions in adolescence by investigating the link between epigenetic changes as an effect of psychotherapy. It investigates the correlation between changes in the methylation of the FKBP5 gene and psychotherapy induced changes in symptoms and functioning.

ELIGIBILITY:
Inclusion Criteria:

* adolescents presenting 3 or more criteria for BPD in the Structured clinical interview for the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) axis II personality disorders (SCID-II)

Exclusion Criteria:

* difficulties to understand or comply with instructions
* psychotic disorders
* pervasive developmental disorders
* severe somatic or neurological disorders
* severe and persistent substance addiction
* elevated risk for complications related to blood sampling

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients in Basel/ Switzerland will be recruited from the routine clinical practice of the Outpatient Department of the Child and Adolescent Psychiatric Hospital.
  Patients in Santiago/ Chile will be recruited from the Department of Psychiatry and Mental Health, East Campus,Faculty of Medicine, University of Chile.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
change in methylation of the FKBP5 gene | after 6 months from baseline
  change in methylation of the FKBP5 gene

SECONDARY OUTCOMES:
change in methylation of the FKBP5 gene | at month 3 and at month 12 after baseline.
  change in methylation of the FKBP5 gene

CONTACTS AND LOCATIONS:
Overall Officials: Ronan Zimmermann, PhD, Principal Investigator — Kinder- und Jugendpsychiatrische Klinik/Universitäre Psychiatrische Klinken Basel (UPK)